CLINICAL TRIAL: NCT04978038
Title: Fourth Dose of Pfizer mRNA COVID-19 Vaccine in Residents of Long-Term Care Facilities
Brief Title: Fourth Dose of mRNA COVID-19 Vaccine in Residents of LTCFs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mark Loeb (Other)
Responsible Party: Sponsor-Investigator, Mark Loeb, M.D., MSc, Professor, Pathology and Molecular Medicine, and Clinical Epidemiology and Biostatistics, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-COVID19-D3-2021
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV2 Infection; Coronavirus Infection
Keywords: COVID-19; Immunization; Long-term care
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — 2019-nCoV Vaccine mRNA-1273; Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, laboratory staff, safety monitoring committee and research assistants will be blinded. To maintain blinding of the participants, those allocated to the control will receive .5ml Prevnar-13 vaccine to mimic mRNA vaccine. Study vaccine will be administered by unblinded nurses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pfizer-BioNtech mRNA- COVID-19 (Experimental): Eligible participants will be vaccinated with the Pfizer-BioNtech mRNA- COVID-19. A 0.3ml dose of the vaccine will be administered intramuscularly.
  Interventions: Drug: mRNA- COVID-19
- Pneumococcal Prevnar-13 (Active Comparator): Eligible participants will be vaccinated with Pfizer Prevar-13 (pneumococcal vaccine) in a blinded manner such that the vaccination with Pfizer-BioNtech mRNA- COVID-19 will be mimicked. That is, a 0.5ml dose of the vaccine will be administered intramuscularly. After completion of the study participants in the control arm will be given a fourth dose of Pfizer-BioNtech mRNA- COVID-19.
  Interventions: Drug: Prevnar13

INTERVENTIONS:
Drug: mRNA- COVID-19 — Pfizer-BioNtech mRNA- COVID-19 0.3ml dose administered intramuscularly
  Other Names: Pfizer-BioNtech mRNA- COVID-19
  Arms: Pfizer-BioNtech mRNA- COVID-19
Drug: Prevnar13 — Pfizer Prevnar-13 pneumococcal vaccine 0.5ml dose administered intramuscularly
  Other Names: Pneumococcal Vaccine
  Arms: Pneumococcal Prevnar-13

SUMMARY:
This study is a multi-centre, blinded, randomized controlled trial. LTCF residents ≥ 65 years who have received three doses of mRNA vaccine will be randomized to vaccination with a fourth dose of Pfizer-BioNtech mRNA- COVID-19 vaccine or to vaccination with a control (Prevnar-13 vaccine).

DETAILED DESCRIPTION:
The primary objective of this study is to test whether vaccinating LTCF residents ≥65 years with a fourth dose of Pfizer-BioNtech mRNA- COVID-19 vaccine as compared to control (PCV13) leads to an increase in detectable neutralizing antibodies. Participants will be randomized to receive either the Pfizer COVID-19 vaccine or the Pnemoccocal Prevnar-13 vaccine at baseline after bloodwork is drawn. Another blood sample will be taken 28 days later. After completion of the study, participants in the control group (pneumococcal Prevnar-13 vaccine) will be given a fourth dose of mRNA COVID-19 vaccine and will have their blood drawn 28 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* LTCF residents ≥ 65 years who have received three doses of mRNA vaccine.

Exclusion Criteria:

* Immunocompromised individuals due to known or suspected immunodeficiency or due to receipt of immunosuppressive medication (e.g., steroids, biologics).
* Having had a severe adverse reaction (e.g., anaphylactic allergy) to mRNA or pneumococcal vaccine.
* Having received pneumococcal polysaccharide vaccine within 12 months.
* LTCF residents who have an interval less than 3 months from their third mRNA COVID vaccine dose.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of neutralizing antibodies | 28 days
  The primary outcome of this study will be detectable neutralizing antibody to the Omicron strain of SARS-CoV-2.

SECONDARY OUTCOMES:
Total IgG spike response | 28 Days
  Secondary Outcome measured using in-house assay for IgG spike protein response
Total IgM spike response | 28 Days
  Secondary Outcome measured using in-house assay for IgM spike protein response
IgA spike antibodies titre | 28 Days
  Secondary Outcome measured using in-house assay for IgA spike protein titre
Anti-RBD antibody titre | 28 Days
  Secondary Outcome measured using in-house assay for Anti-RBD antibody titre
ADCC Response | 28 Days
  Secondary Outcome measured using in-house assay for ADCC response

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Personal identification information removed and assigned a number. Information linked ID to identifying information stored securely at McMaster. Only vaccine administration will have access to identifying information. No personal identification will be published.